CLINICAL TRIAL: NCT04935008
Title: Evaluation of Intracranial Pressure Change by Measuring Optic Nerve Sheath Diameter During Lung Recruitment Maneuver in Patients With Acute Respiratory Distress Syndrome: A Prospective Experimental Study
Brief Title: Evaluation of Intracranial Pressure During Mechanical Ventilation Recruitment Maneuver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ozgur Komurcu, Assistant professor, Ondokuz Mayıs University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/528
Record Dates: First submitted 2021-06-10; First posted 2021-06-22 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Effect of Recruitment Maneuver on Intracranial Pressure
Keywords: Recruitment maneuver; Intracranial pressure; Optic Nerve Sheath Diameter; Acute respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: all patients in mechanical ventilation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effect of recruitment maneuver on intracranial pressure (Experimental): A recruitment maneuver will be performed in patients with decreased oxygen saturation due to atelectasis by applying 30 cm H2O positive pressure support for 30 seconds. The effect of the recruitment maneuver on intracranial pressure will be investigated by measuring the optic nerve sheath diameter with the help of ultrasonography before and after the recruitment maneuver.
  Interventions: Diagnostic Test: The recruitment maneuver

INTERVENTIONS:
Diagnostic Test: The recruitment maneuver — In patients with ARDS, 30 cm H2O positive pressure support and 30 seconds recruitment maneuver will be applied. The effect of the recruitment maneuver on intracranial pressure will be investigated by measuring the optic nerve sheath diameter with the help of ultrasonography before and after the recruitment maneuver. Optic nerve diameter will be evaluated with a linear probe on the eyeball before and after the collection maneuver, taking a value of 3 mm from the eyeball.
  Other Names: Measurement of optic nerve sheath diameter with the help of ultrasonography

SUMMARY:
Recruitment maneuver is used to reopen atelectasis alveoli. Positive airway pressure applied during the recruitment maneuver may increase intrathoracic pressure, resulting in hemodynamic instability, venous return disorders, and increased intracranial pressure. Our study will examine the effect of recruitment maneuver on intracranial pressure by evaluating Optic Nerve Sheath Diameter change.

DETAILED DESCRIPTION:
The therapeutic goal of mechanical ventilation shifts from maintaining regular gas exchange to preventing ventilator-induced lung injury. Atelectasis aggravates lung injury by reducing the lung size available for tidal ventilation. By preventing atelectasis with Positive End Expiratory Pressure (PEEP) and recruitment maneuvers, the end-expiratory lung volume can be increased, and lung damage can be reduced.

Although the recruitment maneuver improves oxygenation and reduces mortality, especially in patients with Acute Respiratory Distress Syndrome (ARDS), adverse side effects are sometimes observed. Most important of these are the risk of barotrauma after positive airway pressure applications, increased intrathoracic pressure and hemodynamic instability, and increased intracranial pressure risk after venous return disorder.

Our study aimed to evaluate the effect of recruitment maneuver on intracranial pressure by measuring optic nerve diameter with ultrasound before and after its application in patients with ARDS with impaired oxygenation and followed up with mechanical ventilator support.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients followed in the Intensive Care Unit (ICU)
* Patients on mechanical ventilation support
* Patients diagnosed with ARDS according to the Berlin criteria
* Patients with oxygen saturation (SpO2) ≤ 92%

Exclusion Criteria:

* Younger than 18
* Patients with increased inotropic drug requirement or mean arterial pressure <65 mmHg in the last 2 hours
* Patients with intracranial hypertension
* Patients with acute coronary syndrome
* Patients with hypercapnia, pneumothorax, subcutaneous emphysema, and pneumomediastinum

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Effect of recruitment maneuver on optic nerve sheath diameter (ONSD) | 1 minute
  Change in optic nerve sheath diameter (ONSD) after the recruitment maneuver in acute respiratory distress syndrome (ARDS) patients

SECONDARY OUTCOMES:
Effect of recruitment maneuver on respiratory compliance (Cdyn) | 10 minute
  Change in respiratory compliance (Cdyn) after the recruitment maneuver
Effect of recruitment maneuver on oxygen saturation (SpO2) | 10 minute
  Change in oxygen saturation (SpO2) after the recruitment maneuver
The effect of change of respiratory compliance (Cdyn) on optic nerve sheath diameter (ONSD) after the recruitment maneuver | 10 minute
  Effect of respiratory compliance (Cdyn) change on optic nerve sheath diameter (ONSD) change after recruitment maneuver

CONTACTS AND LOCATIONS:
Overall Officials: özgür kömürcü, 1, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs Üniversitesi, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cortes I, Penuelas O, Esteban A. Acute respiratory distress syndrome: evaluation and management. Minerva Anestesiol. 2012 Mar;78(3):343-57. PMID 22357372
- [Background] Dreyfuss D, Saumon G. Ventilator-induced lung injury: lessons from experimental studies. Am J Respir Crit Care Med. 1998 Jan;157(1):294-323. doi: 10.1164/ajrccm.157.1.9604014. No abstract available. PMID 9445314
- [Background] Gattinoni L, Agostoni A, Pesenti A, Pelizzola A, Rossi GP, Langer M, Vesconi S, Uziel L, Fox U, Longoni F, Kolobow T, Damia G. Treatment of acute respiratory failure with low-frequency positive-pressure ventilation and extracorporeal removal of CO2. Lancet. 1980 Aug 9;2(8189):292-4. doi: 10.1016/s0140-6736(80)90237-8. PMID 6105441
- [Background] Lim SC, Adams AB, Simonson DA, Dries DJ, Broccard AF, Hotchkiss JR, Marini JJ. Intercomparison of recruitment maneuver efficacy in three models of acute lung injury. Crit Care Med. 2004 Dec;32(12):2371-7. doi: 10.1097/01.ccm.0000147445.73344.3a. PMID 15599138
- [Background] Marini JJ. Recruitment by sustained inflation: time for a change. Intensive Care Med. 2011 Oct;37(10):1572-4. doi: 10.1007/s00134-011-2329-7. Epub 2011 Aug 20. No abstract available. PMID 21858521
- [Background] Amato MB, Barbas CS, Medeiros DM, Magaldi RB, Schettino GP, Lorenzi-Filho G, Kairalla RA, Deheinzelin D, Munoz C, Oliveira R, Takagaki TY, Carvalho CR. Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. N Engl J Med. 1998 Feb 5;338(6):347-54. doi: 10.1056/NEJM199802053380602. PMID 9449727
- [Background] Lapinsky SE, Mehta S. Bench-to-bedside review: Recruitment and recruiting maneuvers. Crit Care. 2005 Feb;9(1):60-5. doi: 10.1186/cc2934. Epub 2004 Aug 18. PMID 15693985